CLINICAL TRIAL: NCT04667793
Title: Clinical Study of Neoadjuvant PD-1 Antibody (Toripalimab) Plus Chemotherapy for Locally Advanced Thymic Epithelial Tumor
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Peng Zhang, Director of science and education department, Shanghai Pulmonary Hospital, Shanghai, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ChestMate-001(FK-NEO-TET-001)
Record Dates: First submitted 2020-12-05; First posted 2020-12-16 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-04

CONDITIONS: Thymic Epithelial Tumor
MeSH Terms: conditions — Thymic epithelial tumor | interventions — toripalimab; Drug Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Thymic Epithelial Tumor (Experimental): For thymoma:
  Neoadjuvant treatment stage: Toripalimab 240mg, q3w, i.v., 2-4 cycles; platinum-based chemotherapy (Carboplatin AUC 5, Amycin 50mg/m2, Cyclophosphamide 500mg/m2) q3w, i.v., 2-4 cycles, then receive chest CT evaluation.
  Surgery stage: the patients will receive radical surgery after the neoadjuvant treatment.
  Adjuvant treatment stage: the patients who did not receive 4 cycle therapy will receive 1-2 cycles therapy up to 4 cycles in total, the following therapy is according to the NCCN guidelines.
  For thymic carcinoma:
  Neoadjuvant treatment stage: Toripalimab 240mg, q3w, i.v., 2-4 cycles; platinum-based chemotherapy (Cisplatin 50mg/m2, Paclitaxel 200mg/m2) q3w, i.v., 2-4 cycles, then receive chest CT evaluation.
  Interventions: Drug: Toripalimab + Chemotherapy

INTERVENTIONS:
Drug: Toripalimab + Chemotherapy — Toripalimab: 200mg, q3w, i.v., 2-4 cycles
  Chemotherapy:
  Thymoma: Cisplatin+Amycin+Cyclophosphamide Thymic carcinoma: Carboplatin+Paclitaxel

SUMMARY:
This is a phase II, single-arm, open-label study to evaluate the efficacy and safety of neoadjuvant Toripalimab + chemotherapy followed by radical surgery as first-line treatment in patients with locally advanced thymic epithelial tumor.

ELIGIBILITY:
Inclusion Criteria:

* Thymic epithelial tumor confirmed by needle biopsy;
* No systemic metastasis confirmed by PET-CT;
* Eastern Cooperative Oncology Group (ECOG) performance-status score of 0 or 1.
* At stage III-IVA (masaoka-koga) as identified by chest CT or MRI;
* With the feasibility or anticipated feasibility after neoadjuvant therapy to receive radical surgery;
* Aged 18-75 years;
* At least 1 measurable lesion according to RECIST 1.1;
* Patients with good function of other main organs (liver, kidney, blood system, etc.):

  * ANC count ≥1.5×10^9/L, platelet count ≥100×10^9/L，hemoglobin ≥90 g/L;
  * the international standard ratio of prothrombin time (INR) and prothrombin time (PT) < 1.5 times of upper limit of normal (ULN);
  * partial thromboplastin time (APTT) ≤1.5×ULN;
  * total bilirubin ≤1.5×ULN;
  * alanine aminotransferase (ALT) aspartate aminotransferase (AST) ≤2.5×ULN, or ALT and AST ≤5×ULN in the patients with liver metastatic tumor.
* The child-bearing female must undergo pregnancy test within 7 days before starting the treatment and the result shall be negative. Reliable contraceptive measures, such as intrauterine device, contraceptive pill and condom, shall be adopted during the trial and within 30 days after completion of the trial. The child-bearing male shall use condom for contraception during the trial and within 30 days after completion of the trial;
* The patient shall sign the Informed Consent Form.

Exclusion Criteria:

* Participants who have received any systemic anti-cancer treatment for thymic epithelial tumor, including surgical treatment, local radiotherapy, cytotoxic drug treatment, targeted drug treatment and experimental treatment;
* Administration of any Chinese medicine against cancer before administration of the drug;
* Participants with other cancer (excluding cervical carcinoma in situ, cured basal cell carcinoma, bladder epithelial tumor [including TA and tis]) within five years before the start of this study;
* Participants with any unstable systemic disease (including active infection, uncontrolled hypertension), unstable angina pectoris, angina pectoris starting in the last three months, congestive heart failure (>= NYHA) Grade II), myocardial infarction (6 months before admission), severe arrhythmia requiring drug treatment, liver, kidney or metabolic diseases;
* With activate or suspectable autoimmune disease, or autoimmune paracancer syndrome requiring systemic treatment;
* Antibiotics were used to treat the infection for 4 weeks prior to the start of the trial;
* Participants who were systemically treated with corticosteroids (prednisone or other corticosteroids >10 mg/ day) or other immunosuppressive agents within 2 weeks prior to first administration. In the absence of active autoimmune disease, inhaled or topical corticosteroids and adrenal hormone replacement therapy with a dose of less than 10 mg/ day of prednisone are permitted;
* Participants who are allergic to the test drug or any auxiliary materials;
* Participants with active hepatitis B, hepatitis C or HIV;
* The vaccine was administered within 4 weeks of the start of the trial;
* Participants who have undergone major surgery or severe trauma in other systems within 2 months before the start of this trial;
* Pleural effusion, pericardial effusion or ascites that are not clinically controlled and require pleural puncture or abdominal puncture drainage within 2 weeks before inclusion;
* The patients have active pia meningioma, uncontrolled or untreated brain metastases;
* Pregnant or lactating women;
* Participants suffering from nervous system diseases or mental diseases that cannot cooperate;
* Participated in another therapeutic clinical study;
* Other factors that researchers think it is not suitable for enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-01-31 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Safety: frequency of severe adverse events | up to 5 months
  The frequency of severe adverse events from the participants enrolling to 30 days after the last drug administration or 30 days after surgery or new anti-cancer therapy, which comes first.
Major pathologic response (MPR) | up to 4 months
  MPR is defined as the proportion of participants who have achieved major pathologic response (on routine hematoxylin and eosin staining, tumors with no more than 10% viable tumor cells) in all participants who have completed the neoadjuvant therapy before surgery.

SECONDARY OUTCOMES:
Objective response rate (ORR) | up to 4 months
  It refers to the proportion of patients who have had a complete response or partial response (according to RECIST1.1) as confirmed by CT evaluation after 3 weeks in all patients who have completed the neoadjuvant therapy. Only patients with measurable lesions at baseline will be analyzed.
Disease-free survival (DFS) | up to 60 months
  It refers to the time from radical surgery to relapse or death of a participant due to disease progression. In the case of a patient who still survives at the time of analysis, the latest evaluation date will be used for interpolation (censoring).
Overall survival (OS) | up to 60 months
  It is defined as the time from enrollment to death of participant due to any cause. In the case of a patient who still survives at the time of analysis, the date of last contact will be taken as the censoring date. In the event of a patient with the survival status unknown, the date when the patient is last known to be alive will be used for interpolation (censoring).
Health related quality of life (HRQol) | up to 6 months
  The assessment is made according to the Quality of Life Scale for Lung Cancer Patients (EORTC-QLQ-C30 & LC13, Version 3). EORTC's QLQ-C30 & LC13 (V3.0) is a core scale for lung cancer patients, with a total of 43 items. Among them, Item 29 and 30 are divided into seven grades, which are assigned with 1 to 7 scores according to the answer options. The other items are divided into 4 grades: Not at All, A Little, Quite a Bit, and Very Much, assigned with 1 to 4 scores respectively. The higher score, the worse quality.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided